CLINICAL TRIAL: NCT00997568
Title: Safety of the PET-511BTM Transesophageal Transducer (TEE)
Brief Title: Safety of the PET-511BTM Transesophageal Transducer
Acronym: TEE
Status: Completed | Type: Observational
Sponsor: Toshiba America Medical Systems, Inc. (Industry)
Responsible Party: Terry Schultz, Manager Regulatory Affairs, Toshiba America Medical Systems, Inc.
Other Study IDs: TEE-001
Record Dates: First submitted 2009-10-15; First posted 2009-10-19 (Estimated); Last update posted 2010-08-20 (Estimated); Status verified 2010-08

CONDITIONS: Patient Requiring TEE Procedure by Their Physician
Keywords: transesophageal; transducer; TEE

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- TEE Procedure: Patients who have been scheduled for a TEE procedure by their physician
  Interventions: Device: PET-511BTM

INTERVENTIONS:
Device: PET-511BTM — Transesophageal Transducer
  Other Names: TEE Transducer; TEE Probe

SUMMARY:
The purpose of this study is to demonstrate the safety of the redesigned transesophageal echocardiogram (TEE) transducer as it is inserted and transitioned into the esophagus through the mouth.

DETAILED DESCRIPTION:
The PET-511BTM is a multiplane transesophageal transducer designed for use with Toshiba Diagnostic Ultrasound Systems for the visualization of the heart (and other organs) as a real-time ultrasound image. It is inserted into the esophagus through the mouth to visualize a plane of the heart through the esophageal wall.

The objective of the study is to demonstrate the safe use of the redesigned Toshibal TEE transducer for ease of passage and during transitioning into and down the esophagus to complete a normal TEE study.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients between the ages of 20 and 80
* Informed consent understood and signed
* Compliance with post-treatment follow-up protocol requirements

Exclusion Criteria:

* None

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who have been scheduled for a TEE procedure by their physician.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2009-10

PRIMARY OUTCOMES:
The TEE transducer passes safely into the esophagus. | during, 30 minutes, and 24 hours after the exam

CONTACTS AND LOCATIONS:
Overall Officials: Gregory B. Clarke, M.D, Principal Investigator — The Christ Hospital; David Rubensen, M.D., Principal Investigator — Scripps Health
Locations (2):
- United States (2):
  - Scripps Health, La Jolla, California
  - The Christ Hospital, Cincinnati, Ohio